CLINICAL TRIAL: NCT02830932
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Determine the Safety and Immunogenicity of an Adenoviral-Vector Based Respiratory Syncytial Virus (RSV) F Protein Vaccine (VXA-RSV-f) Expressing Protein F and dsRNA Adjuvant Administered Orally to Healthy Volunteers
Brief Title: Dose-Ranging Trial of Safety & Immunogenicity of an Oral Adenoviral-Vector Based RSV Vaccine (VXA-RSV-f)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA-RSV-101
Record Dates: First submitted 2016-03-23; First posted 2016-07-13 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VXA-RSV-f Tablets (high dose) (Experimental): Singe dose of orally administered VXA-RSV-f Tablets (high dose). VXA-RSV-f is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of respiratory illness caused by RSV. The vaccine vector encodes for a full-length F protein gene from RSV.
  Interventions: Biological: VXA-RSV-f Tablets (high dose)
- VXA-RSV-f Tablets (low dose) (Experimental): Singe dose of VXA-RSV-f Tablets (low dose).VXA-RSV-f is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of respiratory illness caused by RSV. The vaccine vector encodes for a full-length F protein gene from RSV.
  Interventions: Biological: VXA-RSV-f Tablets (low dose)
- VXA Placebo Tablets (Placebo Comparator): Singe dose of matching placebo tablets. The placebo tablets are small off-white tablets that are similar in size and number to the active vaccine dose being delivered.
  Interventions: Other: VXA Placebo Tablets

INTERVENTIONS:
Biological: VXA-RSV-f Tablets (high dose) — The drug product will be provided as small white enteric-coated tablets. Multiple tablets may be administered to delivered the high dose.
  Other Names: RSV (high dose) Oral Vaccine Tablet
  Arms: VXA-RSV-f Tablets (high dose)
Other: VXA Placebo Tablets — The placebo will be provided as small white enteric-coated tablets that are similar in size and number to the active drug product tablets.
  Other Names: Placebo Control
  Arms: VXA Placebo Tablets
Biological: VXA-RSV-f Tablets (low dose) — The drug product will be provided as small white enteric-coated tablets. Multiple tablets may be administered to delivered the low dose
  Other Names: RSV (low dose) Oral Vaccine Tablet
  Arms: VXA-RSV-f Tablets (low dose)

SUMMARY:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Determine the Safety and Immunogenicity of an Adenoviral-Vector Based Respiratory Syncytial Virus (RSV) F Protein Vaccine (VXA-RSV-f) Expressing Protein F and dsRNA Adjuvant Administered Orally to Healthy Volunteers

DETAILED DESCRIPTION:
The study will enroll 66 subjects in four cohorts. All subjects will receive a single administration of VXA-RSV-f at a low dose, a high dose or placebo.

Two sentinel groups will enroll 3 subjects each in an open-label manner (Cohorts 1 and 3) to receive VXA-RSV-f prior to enrolling either of the randomized, controlled cohorts (Cohorts 2 and 4). Within the double-blinded Cohorts (2 and 4), placebo subjects will receive the same number of tablets as the vaccine subjects in that Cohort. Subjects will be enrolled and dosed in the low dose groups prior to initiation of dosing in the high dose group.

Cohort 1: 3 subjects at low dose Cohort 2: 20 subjects at low dose and 10 placebo Cohort 3: 3 subjects at high dose Cohort 4: 20 subjects at low dose and 10 placebo

Subjects will be followed for 28 days post vaccination for preliminary immunogenicity. Subjects will continue to be followed for 1 year post-vaccination for long term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18 - 49 years, inclusive
2. Able to give written informed consent
3. Healthy (no clinically significant health concerns)
4. Safety laboratory values within the following range criteria normal range
5. Body mass index between 17 and 35 at screening

Exclusion Criteria:

1. Receipt of any investigational RSV vaccine within two years prior to study
2. Receipt of any investigational vaccine, drug or device within 8 weeks preceding vaccination
3. Administration of any licensed vaccine within 30 days prior to study
4. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed at baseline
5. History of drug, alcohol or chemical abuse within 1 year prior to vaccination
6. Presence of a fever ≥ 38oC measured orally at baseline
7. Stool sample with occult blood at screening

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Systemic Reactogenicity of VXA-RSV-f vaccine delivered by oral enteric tablet. | Day 7
  Number of Patients with Systemic Reactogenicity Symptoms

SECONDARY OUTCOMES:
Immunogenicity of VXA-RSV-f vaccine delivered by oral enteric tablet. | Day 28
  Number of Patients with a >/= 4-fold Increase in Serum Neutralizing Antibodies from Baseline as determined by PRNT Assay
Immunogenicity of VXA-RSV-f vaccine delivered by oral enteric tablet (GMT) | Days 7 and 28
  Mean Geometric Mean Titer
Immunogenicity of VXA-RSV-f vaccine delivered by oral enteric tablet (GMFR) | Days 7 and 28
  Mean Geometric Mean Fold Rise

CONTACTS AND LOCATIONS:
Locations (1):
- Optimal Research, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be made available to subjects following the 1 year safety follow-up period.